CLINICAL TRIAL: NCT04242823
Title: Performance of Two-stage Cervical Cancer Screening Algorithms Using Primary High-risk Human Papillomavirus Testing in Botswana
Brief Title: Primary HPV-based Cervical Cancer Screening Algorithms in Botswana
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Botswana (Other); Botswana Harvard AIDS Institute Partnership (Other)
Responsible Party: Principal Investigator, Rebecca Luckett, Obstetrician Gynecologist, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P001130
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline screening cohort (Other): This group undergoes HPV testing using self-collected swabs. Triage evaluation occurs in all women who test HPV positive which includes visual inspection with acetic acid and colposcopy. The WLHIV in the cohort who test HPV positive at baseline but who have concurrent benign histopathology results will be invited back for re-screening at a 2-year interval, and undergo similar HPV testing and triage procedures. The WLHIV in the cohort who test HPV negative at baseline will be invited back for re-screening at a 3-year interval and undergo similar HPV testing and triage procedures.
  Interventions: Diagnostic Test: 8-type HPV genotype restriction

INTERVENTIONS:
Diagnostic Test: 8-type HPV genotype restriction — Participants will undergo primary hrHPV testing and if positive will be referred for VIA per Botswana and WHO guidelines. Participants will also undergo colposcopy and biopsy at the time of VIA. The performance of triage with 8-type HPV genotype restriction will be evaluated.

SUMMARY:
Primary high-risk human papillomavirus (HPV) testing has become first line screening for cervical cancer in high-income countries. The feasibility of this approach in low- and middle-income countries (LMICs) is less clear, as is the role of HPV testing among women living with human immunodeficiency virus (HIV). The proposed study seeks to evaluate the accuracy of cervical cancer screening algorithms using primary HPV testing followed by various forms of visual evaluation, including visual inspection with acetic acid (VIA), colposcopy and automated visual evaluation (AVE) for the detection of high-grade cervical dysplasia, using histology as the gold standard. We will validate the AmpFire Assay for HPV self-sampling in our setting. We will determine safe screening intervals in women living with HIV (WLHIV) in an HPV-based cervical cancer screening program and compare triage strategies for positive HPV results at WHO recommended screening intervals for WLHIV. We also seek to understand in-depth the attitudes, acceptability and preferences regarding cervical cancer screening, HPV testing, and self-sampling, for women in Botswana through interviews of a sub-set of women recruited for the cervical cancer screening study. Finally, we will analyze the cost of two-stage cervical cancer screening algorithms using high-risk HPV testing in Botswana.

ELIGIBILITY:
Inclusion Criteria:

1. Cis-gender female or transgender male (must have a cervix)
2. ≥25 years of age
3. Competent to understand study procedures and give informed consent.

Exclusion Criteria:

1. Currently pregnant (as diagnostic procedures for cervical cancer are often deferred during pregnancy)
2. Previous hysterectomy
3. Previous diagnosis of cervical cancer

Ages: 25 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender female or transgender male are eligible if they have a cervix.
Enrollment: 3000 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Compare the sensitivity, specificity, PPV and NPV of triage of primary human papillomavirus testing with 8-type HPV genotype restriction to visual inspection with acetic acid and colposcopy | 3 years
Determine the persistence of HPV infection in WLHIV at the pre-specified follow-up interval | 5 years
Determine the clearance of HPV infection in WLHIV at the pre-specified follow-up interval | 5 years
Determine the incidence of HPV infection in WLHIV at the pre-specified follow-up interval | 5 years
Quantify the incidence of cervical intraepithelial lesion grade 3 or worse in women living with HIV who were baseline HPV positive but with benign pathology at 2 year interval screening | 5 years
Quantify the incidence of cervical intraepithelial lesion grade 3 or worse in women living with HIV who were baseline HPV negative at 3 year interval screening | 5 years
Analyze the cost of two-stage cervical cancer screening algorithms using high-risk HPV testing in Botswana. | 5 years

SECONDARY OUTCOMES:
Understand in-depth the attitudes, acceptability and preferences regarding cervical cancer screening, HPV testing, and self-sampling, for women in Botswana through interviews of a sub-set of women recruited for the cervical cancer screening study. | 6 years
Evaluate the performance of a novel HPV assay as a stand-alone screening tool in our high-prevalence HIV population | 3 years
Evaluate the impact of patient demographic and clinical factors, such as number of sexual partners, smoking, HIV status and related HIV immune markers, on risk of cervical dysplasia | 5 years
Evaluate the impact of patient characteristics and and risk factors on the risk for cervical disease | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Bamalete Lutheran Hospital, Ramotswa, Botswana

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.

REFERENCES:
- [Derived] Luckett R, Zhang BX, Gompers A, George J, Modest A, Bazzett-Matabele L, Vuylsteke P, Kula M, Monare B, Botha MH, Shapiro RL, Ramogola-Masire D, Grover S. High-grade cervical disease and cervical cancer in women aged 50 years and older compared with younger women: examining prevalence by HIV status in two large prospective cohorts in Botswana. BMJ Open. 2024 Oct 29;14(10):e089375. doi: 10.1136/bmjopen-2024-089375. PMID 39477271
- [Derived] Luckett R, Ramogola-Masire D, Gompers A, Moraka N, Moyo S, Sedabadi L, Tawe L, Kashamba T, Gaborone K, Mathoma A, Noubary F, Kula M, Grover S, Dreyer G, Botha MH, Makhema J, Shapiro R, Hacker MR. Triage of HPV positivity in a high HIV prevalence setting: A prospective cohort study comparing visual triage methods and HPV genotype restriction in Botswana. Int J Gynaecol Obstet. 2024 May;165(2):507-518. doi: 10.1002/ijgo.15225. Epub 2023 Nov 10. PMID 37950533